CLINICAL TRIAL: NCT03463616
Title: MRI Imaging or CT Abdomen as Standard Work-up Before Treatment Planning for Rectal Cancer?
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Mattias Prytz, Principal Investigator, Sahlgrenska University Hospital
Other Study IDs: MRvsCT
Record Dates: First submitted 2018-02-28; First posted 2018-03-13 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Rectal Cancer; Liver Metastases
Keywords: Rectal Cancer; Liver Metastases; CT abdomen; MRI Liver
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CT abdomen: Patients who had a CT abdomen as primary work-up before treatment planning for rectal cancer.
  Interventions: Radiation: CT abdomen
- MRI Abdomen: Patients who had a MRI abdomen as primary work-up before treatment planning for rectal cancer.
  Interventions: Radiation: MRI abdomen

INTERVENTIONS:
Radiation: CT abdomen — CT scan of abdomen for metastasis staging of rectal cancer
  Groups: CT abdomen
Radiation: MRI abdomen — MRI of abdomen for metastasis staging of rectal cancer
  Groups: MRI Abdomen

SUMMARY:
Rectal cancer is a common diagnosis. The prognosis after treatment has improved over the last decades, partly due to neoadjuvant radio(chemo)therapy, but also due to improved surgical technique (TME) and, in certain cases, due to adjuvant therapy after surgery. For some 15-20 years, treatment of metastasis has changed; liver- and lung metastasis in certain situations are surgically removed, or in the liver, treated with ablation (radio-frequency). During the same period the possibilities for chemotherapy of metastatic disease have improved, with new drugs and more drug regimens.

These changes in treatment pathways have required changes in how patients with newly diagnosed rectal cancer are "worked up" pre-treatment. Starting in the early 2000s magnetic resonance imaging of the pelvic area has developed and is today mandatory to be able to adequately stage the tumour and plan for the multi-modal treatment before and after surgery.

In many hospitals the set-up is a combination of computed tomography of the abdomen and chest and to this a MRI of the pelvic organs is added, whereas others have adopted MRI also for the abdominal part, thus having an MRI of the liver for the diagnosis of liver metastasis initially, before surgery. For the chest organs, CT is still normative.

MRI has a higher sensitivity and specificity to detect liver metastasis, compared with CT. In order to plan the liver surgery/ablations, most liver surgeons rely on MRI for detailed information about the position of the metastasis and the relation to large vessels.

The aim of this study is to examine the possible differences in percentage of patients requiring further radiology examinations after basic set-up comparing the routine of initial MRI of abdomen (and pelvic organs) with the routine of initial CT of the abdomen (and MRI of the pelvic organs). Further included is an analysis of the rate of liver metastasis using the two different routines, and finally outcome over 12 months in terms of liver treatment for metastasis.

DETAILED DESCRIPTION:
Background:

Rectal cancer is a common diagnosis in both men and women, more commonly occurring in men (60%) than women (40%). In Sweden some 2000 cases are diagnosed each year. The prognosis after treatment has improved over the last decades, partly due to neoadjuvant radio(chemo)therapy, but also due to improved surgical technique (TME) and, in certain cases, due to adjuvant therapy after surgery.

For some 15-20 years, treatment of metastasis has changed; liver- and lung metastasis in certain situations are surgically removed, or in the liver, treated with ablation (radio frequency). During the same period the possibilities for chemotherapy of metastatic disease have improved, with new drugs and more drug regimens.

These changes in treatment pathways have required changes in how patients with newly diagnosed rectal cancer are "worked up" pre-treatment. Starting in the early 2000s magnetic resonance imaging of the pelvic area has developed and is today mandatory to be able to adequately stage the tumour and plan for the multi-modal treatment before and after surgery.

In many hospitals the set-up is a combination of computed tomography of the abdomen and chest and to this a MRI of the pelvic organs is added, whereas others have adopted MRI also for the abdominal part, thus having an MRI of the liver for the diagnosis of liver metastasis initially, before surgery. For the chest organs, CT is still normative.

MRI has a higher sensitivity and specificity to detect liver metastasis, compared with CT. In order to plan the liver surgery/ablations, most liver surgeons rely on MRI for detailed information about the position of the metastasis and the relation to large vessels.

The objective of the study is to examine:

The possible differences in percentage of patients requiring further radiology examinations after basic set-up comparing the routine of initial MRI of abdomen (and pelvic organs) with the routine of initial CT of the abdomen (and MRI of the pelvic organs). Further included is an analysis of the rate of liver metastasis using the two different routines, and finally outcome over 12 months in terms of liver treatment for metastasis.

Hypothesis:

Primary:

• Patients who underwent initial abdominal MRI had a significantly lower need for additional radiology examinations compared with those who underwent initial CT abdomen.

Secondary:

* A higher proportion of patients who underwent initial abdominal MRI underwent liver treatment aiming for cure at 12 months.
* Abdominal MRI as initial examination resulted in a higher proportion of detected liver metastasis.
* Cost effectiveness analysis will show that initial abdominal MRI of the abdominal organs is cost-effective.

Design:

A retrospective study using clinical details such as date for diagnosis, clinical tumour stage, type of surgical treatment and date, pathology tumour stage, local recurrence and survival at 36 months from the Swedish ColoRectal Cancer Registry for patients with rectal cancer treated at Sahlgrenska University Hospital and Norra Älvsborg Hospital during the years collecting patients backwards from 2015-12-31 until sufficient number is reached (see below "Sample size").

Data will be collected in the radiology patient documentation at the two hospitals using the original radiology report for the index examinations as well as type and number of additional radiology examinations and the reports for those.

For patients with liver metastases in the original radiology report at the index work-up and in cases with indeterminate initial results, the original radiology examinations will be re-evaluated by one or if possible two radiologists.

Data from the clinical patient records on treatment plan (index treatment) and time and type of treatment for liver metastasis.

No direct contact with patients is planned, and only data already collected (see above) will be used.

Methodology:

Through Regional Cancer Center West (RCC Väst) appropriate data from to Swedish ColoRectal Cancer Register will be collected, consisting of age, time for diagnosis, time for multidisciplinary conference, time for oncological treatment, time for surgery, cTNM as well as pTNM, performed treatment/s within 12 months, recurrence/s and survival (3 years).

Data to be collected from radiology reports include presence of liver metastasis, number of liver metastasis, additional radiology examinations after index work-up - type and number as well as findings of liver metastasis. Additional findings of distant metastases to retro peritoneal lymph-nodes and to peritoneum will also be recorded.

Data from re-evaluation of examinations for all patients diagnosed with liver metastases such as number of metastases, number of small metastases (<10mm), metastases to retro peritoneal lymph-nodes and to peritoneum.

Data to be collected from hospital records for all patients include time line for different aspects of treatment including multidisciplinary conference (and decision), oncological treatment and liver surgery until 12 months from diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* All patients in the Swedish Colo- Rectal Cancer Registry (SCRCR) and treated for rectal cancer at Sahlgrenska University Hospital and Norra Älvsborg Hospital 2013-2015.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients in the Swedish Colo- Rectal Cancer Registry (SCRCR) and treated for rectal cancer at Sahlgrenska University Hospital and Norra Älvsborg Hospital 2013-2015.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who needed additional radiology examination/s before treatment planning after routine MRI of abdominal organs compared with routine CT of abdominal organs. | 3 months

SECONDARY OUTCOMES:
Comparison of percentage of patients treated with liver surgery/ablation within 12 months between the two groups. | 12 months
Comparison of the percentage of patients who were diagnosed with liver metastasis, between the two groups. | 3 years
Cost effectiveness analysis of routine MRI of abdominal organs compared with routine CT of abdominal organs. | 3 years
  Total cost differences between MRI and CT-scan as primary routine work-up measured in USD.
Overall survival after 3 years | 3 years
Disease free survival after 3 years | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Prytz, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska university hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Park J, Block M, Bock D, Kalebo P, Nilsson P, Prytz M, Haglind E. A Comparison of Liver MRI and Contrast-Enhanced CT as Standard Workup Before Treatment for Rectal Cancer in Usual Care - A Retrospective Study. Curr Med Imaging. 2022;18(2):256-262. doi: 10.2174/1573405617666210712125028. PMID 34931986